CLINICAL TRIAL: NCT04209322
Title: Trial of Pulsed Radiofrequency for Sciatica and Disc Herniation
Acronym: PRATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, Associated Professor of Radiology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF003
Record Dates: First submitted 2019-12-10; First posted 2019-12-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Sciatica; Lumbar Disc Herniation
Keywords: sciatica; lumbar disc herniation; radiofrequency; non invasive treatment
MeSH Terms: conditions — Sciatica; Intervertebral Disc Displacement | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, randomized trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Radiofrequency (Experimental): Aseptic technique was adopted. Imaging guided (CT) catheter needle (active tip electrode) was inserted and a sensory stimulation test was carried out using an RF generator. The catheter needle was then advanced toward the DRG until the patient reported a tingling sensation and/or dysesthesia at less than 0.3V. PRF treatment was administered at 5 Hz and a 2 ms pulsed width for 10 minutes at 45V under the constraint that the electrode tip temperature not exceed 42°C. Finally, patients received 1mL lidocaine 20mg/mL mixed with 2mL dexamethasone 10mg/mL.
  Interventions: Procedure: pulsed Radiofrequency
- Transforaminal Epidural Steroid Injection (Active Comparator): Aseptic technique was adopted. Imaging guided (CT) catheter needle (active tip electrode) was inserted and a sensory stimulation test was carried out using an RF generator. The catheter needle was then advanced toward the DRG until the patient reported a tingling sensation and/or dysesthesia at less than 0.3V. After 10 minutes await (as per pRF), patients received 1mL lidocaine 20mg/mL mixed with 2mL dexamethasone 10mg/mL.
  Interventions: Procedure: Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: pulsed Radiofrequency — Non-surgical treatment of lumbar disc herniation causing sciatica using pulsed radiofrequency (10 minutes) directed to the interested dorsal root ganglia (percutaneous technique); after radiofrequency application, using the same needle, steroid was administered (as per the control arm). The procedure was guided by CT imaging
  Arms: Pulsed Radiofrequency
Procedure: Transforaminal Epidural Steroid Injection — Percutaneous injection of steroid in the nerve root foramen. The procedure was guided by CT imaging
  Arms: Transforaminal Epidural Steroid Injection

SUMMARY:
Transforaminal epidural injection of treatments, commonly steroids (TFESI), is offered to people with sciatica and might improve symptoms, reduce disability and speed up return to normal activities (NICE guidelines) Imaging-guided TFESI has traditionally been performed in the sciatica context because injection is administered directly to the nerve root, which relieves the pain markedly; however, the maintenance time is usually short.

Treatment with radiofrequency for pain management is in clinical use since decades primarily with nerve lesioning (thermoablation) once the specific pain tributary nerve is identified.

Pulsed radiofrequency (PRF) with neuromodulation intention (not lesioning) has been shown to be effective in reducing some types of chronic pain, both degenerative and neuropathic.

Pulsed radiofrequency has been also extensively used in the context of acute and subacute sciatica due to disc herniation without sufficient level of evidence. In a prospective RCT, comparing prf directed to dorsal root ganglia and Tfesi in patients with sciatica did not allow conclusions on efficacy because of limitations of the trial. In that trial, only few participants completed the study due to violation of trial protocol translating the results as not consistent.

One retrospective trial, in which the use of Prf in addition to tfesi was evaluated in patients with acute and subacute sciatica, demonstrated rapid pain relief onset and prolonged maintenance; the overall efficacy was superior to that of the single method treatment (either tfsei or prf).

The investigators conducted a randomized, double-blind, controlled trial (Pulsed Radiofrequency in Addition to Tfesi for Sciatica [PRATS]) to determine if PRF in addition to TFESI leads to better outcomes in the management of patients with acute and subacute sciatica due to disc herniation, compared to TFESI alone.

DETAILED DESCRIPTION:
The investigators conducted a multicenter, prospective, randomized trial among patients with at least 6 weeks of sciatic pain to determine whether a strategy of PRF in addition to TFESI leads to better outcomes during the first year than does a strategy of TFESI only means for sciatica treatment.

Eligible patients were 18 to 75 years of age, had a radiologically confirmed disk herniation, and had received a diagnosis from an attending neurologist of an incapacitating lumbosacral radicular syndrome that had lasted for at least 12 weeks. Correlation of magnetic resonance imaging (MRI) findings with symptoms was registered. Patients presenting with cauda equina syndrome, muscle paralysis, or insufficient strength to move against gravity were excluded. Other exclusion criteria were cardiac pace-maker implant, pregnancy, or severe coexisting disease. The occurrence of another episode of symptoms similar to those of the current episode during the previous 12 months, previous spine surgery and spondylolisthesis were not considered contraindications but bony stenosis.

A computer-generated permuted-block scheme was used for randomization, with an unstratified variable-block size of 2 and 4. The order of blocks was also randomized with patients assigned (1:1) to PRF/TFESI (treatment) or TFESI (control). A few hours before randomization, the patients were evaluated again, and those who had recovered from their symptoms at that time were excluded from the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients had radiologically confirmed disk herniation, and had received a diagnosis from an attending neurologist of an incapacitating lumbosacral radicular syndrome that had lasted for at least 12 weeks. Correlation of magnetic resonance imaging (MRI) findings with symptoms was required.
* The occurrence of another episode of symptoms similar to those of the current episode during the previous 12 months were not considered contraindications

Exclusion Criteria:

* Patients presenting with previous spine surgery, spondylolisthesis, cauda equina syndrome, muscle paralysis, or insufficient strength to move against gravity were excluded.
* Vertebral canal stenosis
* Other exclusion criteria were cardiac pace-maker implant, pregnancy, or severe coexisting disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Leg-Pain Intensity | 52 weeks
  The primary outcome was the average leg-pain intensity score over the course of the previous 1 week (on a numerical pain-rating scale from 0 to 10, with 0 indicating no pain and 10 the worst possible pain; clinically important difference, 2 points), as assessed at 1 week and 52 weeks.

SECONDARY OUTCOMES:
Roland Morris disability questionnaire | 52 weeks
  extent of disability as measured on the Roland Disability Questionnaire for Sciatica (scores range from 0 to 23, with higher scores indicating greater disability; clinically important difference, 8 points), as assessed at 4 weeks, 12 weeks and 52 weeks.
Oswestry Disability Index questionnaire | 52 weeks
  extent of disability as measured on the Oswestry Disability Index (on a % scale from 0 to 100, version 2.0, MODEMS; clinically important difference, 10 points), as assessed at 4 weeks, 12 weeks and 52 weeks.
Pain change questionnaire | 52 weeks
  global perceived effect (post-treatment symptoms as compared with baseline, on a scale from -5 [vastly worse] to 0 [unchanged], to +5 [completely recovered])

OTHER OUTCOMES:
Adverse events | 52 weeks
  Data regarding treatment-related side-effects will be registered.
workplace absenteeism questionnaire | 52 weeks
  The cumulative number of days of workplace absenteeism due to sciatica
Satisfaction on current condition | 52 weeks
  Subjective evaluation of current condition, expressed in terms of percentage, with 0% indicating completely disappointed and 100% indicating completely satisfied

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro Sana, Aprilia, LT
  - Alessandro Napoli, Rome

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data are available to all authors for 5 years after main study completion